CLINICAL TRIAL: NCT04869878
Title: Inter-rater Reliability of the Clinical Frailty Scale in a Swedish Emergency Department Setting
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Daniel Wilhelms, Principal Investigator, University Hospital, Linkoeping
Other Study IDs: 2021-00875IRR
Record Dates: First submitted 2021-04-26; First posted 2021-05-03 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Frailty
Keywords: Inter-rater reliability; Clinical Frailty Scale; Frailty assessment; Frailty; Observer variation; Emergency service
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frailty is a common clinical syndrome in older adults, which may be assessed through various assessment tools. One frequently used tool is the Clinical Frailty Scale (CFS) which potentially can be adopted for daily use in the Emergency Department and has been appraised for reliability to some extent, but have so far not been evaluated in the Swedish emergency care context.

The purpose of this study is to evaluate the inter-rater reliability of the Clinical Frailty Scale (CFS) in a clinical Swedish Emergency Department (ED) setting. Members of multidisciplinary emergency care teams will conduct the assessments individually.

DETAILED DESCRIPTION:
The CFS is introduced and tested as part of a quality-improvement process regarding elderly people within the Emergency departments (EDs) of Region Östergötland (Östergötland County) in Sweden.

CFS is a 9-point scale developed within the Canadian Study of Health and Aging. It comprises of a pictograms and a clinical description to help assign scores ranging from very fit to terminally ill. CFS enables clinicians to rapidly stratify the degree of frailty in the elderly with the help of questions and clinical assessment. However, since the assessment is judgement based, it is important that the inter-rater reliability is satisfactory.

This study is part of a larger project where all eligible patients who visit the ED (24/7) for a period of four weeks will be enrolled and then subsequently assessed with CFS by one of their responsible health-care professionals (i.e. physician, registered nurse or nurse assistant). For this study, each professional on the team will individually assess each patient. First, a clinical judgement is performed (frail/not frail) without any instrument, and then the patient is assessed by using the CFS. This will take place during work shifts when someone from the research team is present and can arrange the assessments, as well as ensure that they are conducted independently. These work shifts will be selected using the online application Research Randomizer, to randomly include all hours of the day as well as eligible health-care professionals.

The research-team member will collect the assigned CFS-scores and information on the age, gender, profession, position (emergency physician or intern/resident from other specialities) and the number of years in the profession of each assessor. Informed consent will be obtained from all health-care professionals who participate. No data that can identify any patient will be collected.

Sample size is determined to be 100 patients, which would be more than sufficient with a power of 90% and α 0,05.

ELIGIBILITY:
Inclusion Criteria:

Health-care professionals:

- Working in the ED, as part of the emergency-care team that are responsible for a patient ≥65 years

Patients:

- ≥65 years

Exclusion Criteria:

Health care professionals:

- Unwilling to provide informed consent

Patients:

- ≤65 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Health care professionals:
  Physicians, nurses and assistant nurses who are the responsible healthcare professionals for the enrolled patients
  Patients:
  Patients of all genders at the age of ≥65 years seeking medical care at the three ED instances in Region Östergötland.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Level of inter-rater reliability regarding frailty as assessed by CFS | The assessment will be made in connection with the patient´s first meeting with the care team, i.e. within 1 hour from the patient´s arrival to the ED
  Inter-rater reliability of the CFS, expressed as Intraclass Correlation Coefficient

SECONDARY OUTCOMES:
Level of correlation between degree of frailty (CFS 1-9) and degree of inter-rater reliability | The assessment will be made in connection with the patient´s first meeting with the care team, i.e. within 1 hour from the patient´s arrival to the ED
  Investigates whether inter-rater reliability, expressed as Intraclass Correlation Coefficient, varies between scale scores in CFS. Described descriptively.
Agreement between CFS and clinical judgement (frail/not frail) | The clinical judgement is made just before the assessment with CFS
  Investigates the agreement between a clinical judgement (with no frailty tool) regarding the patient being frail or not, compared to frailty according to the CFS (cut-off 5). Expressed as a percentage.

OTHER OUTCOMES:
Difference in measures for Inter-rater reliability, expressed as Intraclass Correlation Coefficient, between care teams with emergency physicians in relation to care teams with interns/residents from other specialties. | The assessment will be made in connection with the patient´s first meeting with the care team, i.e. within 1 hour from the patient´s arrival to the ED
  An Emergency department in Sweden typically has physicians from other specialities who work for a period of time. They may not have the same education and training in CFS assessments, we want to explore if the results differ in terms of inter-rater reliability between care teams with emergency physicians and care teams with other physicians.

CONTACTS AND LOCATIONS:
Locations (1):
- Akutmottagningen US Östergötland, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manfredi G, Midao L, Paul C, Cena C, Duarte M, Costa E. Prevalence of frailty status among the European elderly population: Findings from the Survey of Health, Aging and Retirement in Europe. Geriatr Gerontol Int. 2019 Aug;19(8):723-729. doi: 10.1111/ggi.13689. Epub 2019 May 30. PMID 31146300
- [Background] Collard RM, Boter H, Schoevers RA, Oude Voshaar RC. Prevalence of frailty in community-dwelling older persons: a systematic review. J Am Geriatr Soc. 2012 Aug;60(8):1487-92. doi: 10.1111/j.1532-5415.2012.04054.x. Epub 2012 Aug 6. PMID 22881367
- [Background] Preston L, Chambers D, Campbell F, Cantrell A, Turner J, Goyder E. What evidence is there for the identification and management of frail older people in the emergency department? A systematic mapping review. Southampton (UK): NIHR Journals Library; 2018 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK493681/ PMID 29697231
- [Background] Lewis ET, Dent E, Alkhouri H, Kellett J, Williamson M, Asha S, Holdgate A, Mackenzie J, Winoto L, Fajardo-Pulido D, Ticehurst M, Hillman K, McCarthy S, Elcombe E, Rogers K, Cardona M. Which frailty scale for patients admitted via Emergency Department? A cohort study. Arch Gerontol Geriatr. 2019 Jan-Feb;80:104-114. doi: 10.1016/j.archger.2018.11.002. Epub 2018 Nov 8. PMID 30448693
- [Background] Kaeppeli T, Rueegg M, Dreher-Hummel T, Brabrand M, Kabell-Nissen S, Carpenter CR, Bingisser R, Nickel CH. Validation of the Clinical Frailty Scale for Prediction of Thirty-Day Mortality in the Emergency Department. Ann Emerg Med. 2020 Sep;76(3):291-300. doi: 10.1016/j.annemergmed.2020.03.028. Epub 2020 Apr 24. PMID 32336486
- [Background] Lo AX, Heinemann AW, Gray E, Lindquist LA, Kocherginsky M, Post LA, Dresden SM. Inter-rater Reliability of Clinical Frailty Scores for Older Patients in the Emergency Department. Acad Emerg Med. 2021 Jan;28(1):110-113. doi: 10.1111/acem.13953. Epub 2020 Apr 2. No abstract available. PMID 32141671
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Hallgren KA. Computing Inter-Rater Reliability for Observational Data: An Overview and Tutorial. Tutor Quant Methods Psychol. 2012;8(1):23-34. doi: 10.20982/tqmp.08.1.p023. PMID 22833776
- See also: A simplified guide to determination of sample size requirements for estimating the value of intraclass correlation coefficient — https://www.researchgate.net/publication/318788161_A_simplified_guide_to_determination_of_sample_size_requirements_for_estimating_the_value_of_intraclass_correlation_coefficient_A_review
- See also: Randomizer.org — https://www.randomizer.org/

DOCUMENTS (1):
  • Informed Consent Form (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT04869878/ICF_000.pdf